CLINICAL TRIAL: NCT04262895
Title: TTI-0102, a Cysteamine Precursor for Mild to Moderate TBI: Dosing and Feasibility Study
Brief Title: TTI-0102 for Veterans With TBI
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn due to delay in FDA IND submission
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N3323-P; I21RX003323-01 (NIH)
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Mild to Moderate TBI; Posttraumatic Stress Disorder
Keywords: cognition; neurobehavioral symptoms; psychiatric symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — cysteamine-pantetheine disulfide

STUDY DESIGN:
Intervention Model Description: In Phase 1, the investigators will determine whether TTI-0102 2 mg/day or 4 mg/day is more tolerated and/or more effective compared with placebo in Veterans with mild to moderate TBI and PTSD. In Phase 2, the investigators will determine the feasibility and acceptability of trial procedures involving TTI-0102 (dose determined in Phase 1) vs placebo in Veteran participants receiving Compensatory Cognitive Training.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Doses of drug and placebo will be prepared in identical sachets, with group assignment known only to the research pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- TTI-0102 2 mg/day (Experimental): TTI-0102 2 mg/day
  Interventions: Drug: TTI-0102
- TTI-0102 4 mg/day (Experimental): TTI-0102 4 mg/day
  Interventions: Drug: TTI-0102
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTI-0102 — TTI-0102 is a cysteamine precursor.
  Arms: TTI-0102 2 mg/day; TTI-0102 4 mg/day
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Traumatic brain injury (TBI) is a signature wound of the recent wars. How chronic TBI symptoms develop after a mild brain injury is not fully understood, but it is now thought that injury results in damage that reduces brain energy production, increases inflammation, and results in a leaky blood-brain barrier. Difficulties in daily function may persist in areas such as thinking (e.g., attention, learning, memory, planning, and problem-solving), pain (e.g., headache) and behavior (e.g., sleep, posttraumatic stress disorder, depression). No medications for TBI have been developed, so evidence-based cognitive rehabilitation interventions such as Compensatory Cognitive Training (CCT) are the mainstay of treatment. The investigators are proposing to study a medication, TTI-0102, that shows anti-inflammatory activity, as a potential adjunct treatment with CCT for Veterans with TBI-related symptoms. The investigators plan to first determine the best dose of TTI-0102 to use, and then to conduct a pilot study to test the feasibility and acceptability of combining TTI-0102 with CCT in Veterans with mild to moderate TBI and PTSD.

DETAILED DESCRIPTION:
Approximately 12-23% of returning service members report a history of traumatic brain injury, mostly mild (mTBI). Post-concussive symptoms such as memory problems, irritability, and difficulty concentrating are common after TBI and may become chronic, interfering with successful return to duty or civilian reintegration, reducing quality of life, and increasing health care utilization for Veterans. In those whose TBI-related symptoms persist, there is accumulating evidence for increased morbidity (e.g., worse PTSD symptoms, chronic hypopituitarism, dementia), spurring efforts to improve diagnosis and intervention. Following a primary TBI injury, secondary injury and persistent symptoms may evolve through a complex cascade of events that culminate in inflammation, alterations in mitochondrial bioenergetics, and diminished blood brain barrier integrity, ultimately yielding a chronic disease state. To date, Veterans receiving strategy-based cognitive rehabilitation for TBI (CCT/CogSMART) have shown improvement in cognition and subjective neuropsychiatric symptoms. CCT is an evidence-based cognitive rehabilitation intervention emphasizing training in cognitive strategies to improve post-concussive symptoms, attention, learning/memory, and executive functioning. However, no pharmaceuticals have been developed for direct or adjunct-to CCT use to maximize treatment outcomes.

Given that inflammation has been observed in TBI, PTSD, and in co-occurring TBI/PTSD, it may be an important aspect of the TBI/PTSD disease state that could be manipulated to promote healing. The investigators are proposing to study TTI-0102, a cysteamine precursor that shows anti-inflammatory activity, as a potential adjunct to CCT for Veterans with TBI-related symptoms. TTI-0102 is a safe, easily administered, highly-water soluble compound that readily crosses the blood brain barrier. Compared with cysteamine, TTI-0102 degrades more slowly, dampening peak drug concentrations and sustaining drug plasma concentrations in a narrow therapeutic range. Developed to treat cystinosis, cysteamine is now believed to have potential for treatment of neurodegenerative disorders.

The goal of this proof of concept study is first, in Phase I (Year 1), to use symptom change (i.e., objective cognitive performance and subjective cognitive and neuropsychiatric symptoms) and biological profiles (i.e., metabolomics, inflammatory peptides [interleukin-6 and C-reactive protein], and brain-derived neurotrophic factor) to learn optimal dosing of TTI-0102 and to assess mechanism of action, and in Phase II (Year 2), to implement a feasibility trial in Veterans with a history of mild to moderate TBI and PTSD. In Phase I, 3 groups of 10 Veterans each will be randomly assigned to receive TTI-0102 2 grams/day, 4 grams/day, or placebo for 12 weeks. Baseline and post-treatment measures of objective cognition and subjective cognitive and neuropsychiatric symptoms will be administered, and plasma will be collected to measure the metabolomic, inflammatory, and protein biomarkers. In Phase II (Year 2), 12 different Veterans (6 per group) will be enrolled in a pilot randomized controlled trial (RCT) to assess the feasibility and acceptability of trial procedures. Participants in Phase II will be randomized to receive TTI-0102 (dose determined in Phase I) or placebo for 12 weeks as an adjunct to evidence-based CCT. The results of these double-blind, placebo-controlled trials will be used to plan a larger, fully-powered trial.

ELIGIBILITY:
Inclusion Criteria:

* Veteran receiving care at the VA San Diego Healthcare system
* age 18-65
* history of mild to moderate TBI (loss of consciousness <24 hours; posttraumatic amnesia <7 days)
* documented impairment (>1 standard deviation below the mean) in at least one neuropsychological domain as determined by valid clinical neuropsychological testing using at least one performance validity test, i.e.:

  * attention
  * processing speed
  * working memory
  * learning, memory
  * executive functioning
  * DSM-5 diagnosis of PTSD based on the Clinician-Administered PTSD Scale

Exclusion Criteria:

* current alcohol and/or substance abuse or dependence
* high risk for homicide or suicide
* evidence of a significant uncontrolled/unstable medical illness or clinically significant surgery
* laboratory values that are significantly outside normal limits
* history of intolerance or hypersensitivity to cysteamine or penicillamine
* current participation in other intervention studies
* pregnant or intending to become pregnant in the next 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Objective cognition | Change from 0 to 12 weeks
  Mean z-score of objective cognitive measures (Wechsler Adult Intelligence Scale-4th Edition Digit Span, WAIS-IV Coding, Hopkins Verbal Learning Test-Revised, Brief Visuospatial Memory Test-Revised, Delis-Kaplan Executive Function System Trails, D-KEFS Color-Word Interference, D-KEFS Verbal Fluency)

SECONDARY OUTCOMES:
Subjective cognition | Change from 0 to 12 weeks
  Mean z-score of subjective cognitive measures (Neuro-QOL Applied Cognition Executive Function, Neuro-QOL Applied Cognition General Concerns)
Neuropsychiatric symptoms | Change from 0 to 12 weeks
  Mean z-score of subjective neuropsychiatric symptom measures (Neurobehavioral Symptom Inventory Patient Health Questionnaire-9, General Anxiety Disorder-7, Insomnia Severity Index, PTSD Checklist for DSM-5, WHO Disability Assessment Schedule 2.0)
high-sensitive C-reactive protein | Change from 0 to 12 weeks
  high-sensitive C-reactive protein Plasma high sensitivity C-reactive protein (hsCRP) will be measured using the Quantikine HS ELISA kit. The assay sensitivity is 10 pg/ml, the standard range is linear to 100 pg/ml, and intra- and inter-assay CVs are 4.1% and 6.5%, respectively.
interleukin-6 | change from 0 to 12 weeks
  interleukin-6 Plasma interleukin-6 (IL-6) will be measured using the Quantikine HS ELISA kit. The assay sensitivity is 0.70 pg/ml, the standard range is linear to 100 pg/ml, and intra- and inter-assay CVs are 2.6% and 4.5%, respectively.
brain-derived neurotrophic factor | change from 0 to 12 weeks
  brain-derived neurotrophic factor We will use the Quantikine direct ELISA that selectively detects plasma levels of free brain-derived neurotrophic factor (BNDF) without measuring BDNF bound to blood protein that occurs with ELISAs that detect total BDNF. Specificity of this BDNF immunoassay has been further confirmed by using Western blots to detect BDNF levels in plasma that were also measured with the Quantikine BDNF ELISA. We will use our previously established protocol to increase ELISA sensitivity to <4 pg/ml and maximize performance by blocking nonspecific binding on the 96-well plate and optimizing incubation times and other variables for the Quantikine free BDNF ELISA. The intra- and inter-assay CVs for the BDNF ELISA are 4.4% and 7.8%, respectively.
kynurenine metabolism | change from 0 to 12 weeks
  kynurenine metabolism Kynurenine metabolism will be assessed by broad-spectrum, targeted metabolomics using high performance liquid chromatography-tandem mass spectrometry (LC/MS/MS). Paired samples from each participant will be analyzed comparing baseline and TTI-0102-associated changes.
sphingolipid metabolism | change from 0 to 12 weeks
  sphingolipid metabolism Sphingolipid metabolism will be assessed by broad-spectrum, targeted metabolomics using high performance liquid chromatography-tandem mass spectrometry (LC/MS/MS). Paired samples from each participant will be analyzed comparing baseline and TTI-0102-associated changes.
purine metabolism | change from 0 to 12 weeks
  purine metabolism Purine metabolism will be assessed by broad-spectrum, targeted metabolomics using high performance liquid chromatography-tandem mass spectrometry (LC/MS/MS). Paired samples from each participant will be analyzed comparing baseline and TTI-0102-associated changes.
eicosanoid metabolism | change from 0 to 12 weeks
  eicosanoid metabolism Eicosanoid metabolism will be assessed by broad-spectrum, targeted metabolomics using high performance liquid chromatography-tandem mass spectrometry (LC/MS/MS). Paired samples from each participant will be analyzed comparing baseline and TTI-0102-associated changes.
sulfur amino acid metabolism | change from 0 to 12 weeks
  sulfur amino acid metabolism Sulfur amino acid metabolism will be assessed by broad-spectrum, targeted metabolomics using high performance liquid chromatography-tandem mass spectrometry (LC/MS/MS). Paired samples from each participant will be analyzed comparing baseline and TTI-0102-associated changes.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W. Twamley, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study completion, indefinitely.
Access Criteria: Upon request.